CLINICAL TRIAL: NCT04706468
Title: A Phase 2, Multicenter, Randomized, Double-blind, Dose-ranging Study to Evaluate the Efficacy and Safety of TG-1000 Compared With Placebo in Adult Patients With Acute Uncomplicated Influenza Virus Infection
Brief Title: To Evaluate the Efficacy and Safety of TG-1000 Compared With Placebo in Adult Patients With Acute Uncomplicated Influenza Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG-1000-C-02
Record Dates: First submitted 2021-01-06; First posted 2021-01-12 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Influenza Virus Infection

STUDY DESIGN:
Intervention Model Description: A Phase 2, Multicenter, Randomized, Double-blind, Dose-ranging
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 40 mg TG-1000 (Experimental): Participants received 40 mg of TG-1000 and 40 mg of placebo orally on Day 1 and 40 mg of placebo on Day 3.
  Interventions: Drug: TG-1000
- 80 mg TG-1000 (Experimental): Participants received 80 mg of TG-1000 orally on Day 1 and 40 mg of placebo on Day 3.
  Interventions: Drug: TG-1000
- 40 mg TG-1000+40 mg TG-1000 (Experimental): Participants received 40 mg of TG-1000 and 40 mg of placebo orally on Day 1 and 40 mg of TG-1000 on Day 3.
  Interventions: Drug: TG-1000
- Placebo (Placebo Comparator): Participants received 80 mg of placebo orally on Day 1 and 40 mg of placebo on Day 3.
  Interventions: Drug: TG-1000

INTERVENTIONS:
Drug: TG-1000 — Capsules taken orally

SUMMARY:
To evaluate the antiviral effect of TG-1000 compared with placebo in adult patients with acute uncomplicated influenza virus infection.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, dose-ranging study to evaluate the efficacy and safety of different doses of TG-1000 compared with placebo in adult patients with acute uncomplicated influenza virus infection.

Approximately 200 patients will be randomly assigned to 1 of 4 treatments groups in a ratio of 1:1:1:1 to receive study treatment orally: "40 mg TG-1000", "80 mg TG-1000", "40mg+40mg TG-1000" or "placebo".

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Age ≥ 18 (or legal adult age) to < 65 years at the time of signing the informed consent.
3. Must have a positive result of Rapid influenza diagnostic test (RIDT) or Polymerase chain reaction (PCR).
4. The time interval between the onset of symptoms and the randomization is 48 hours or less.
5. Must be able to comply with all study procedures and assessments, including completion of the patient diary.

Exclusion Criteria:

1. Patients with severe influenza virus infection requiring inpatient treatment.
2. Patients with high risk factors may develop into severe cases.
3. Investigator suspects or confirms that patients with bronchitis, pneumonia, pleural effusion or interstitial disease through chest imaging examination.
4. Acute respiratory infection, otitis media or sinusitis within 2 weeks prior to Screening.
5. Purulent sputum or purulent tonsillitis.
6. Positive nucleic acid test for COVID-19.
7. Suspects allergic to active ingredients or excipients.
8. Body weight < 40 kg.
9. Has received anti-influenza drug.
10. Has received any investigational agents or devices for any indication within 30 days prior to Screening.
11. Patients who, in the opinion of the Investigator, may not be qualified or suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
The antiviral effect of TG-1000 compared with placebo in adult patients with acute uncomplicated influenza virus infection. | Up to Day 9
  The time between the initiation of the study treatment and the first time when the influenza virus RNA cannot be detected.

SECONDARY OUTCOMES:
Time to alleviation of all influenza symptoms. | Up to Day 9
  The time between the initiation of the study treatment and the alleviation of influenza symptoms.
The percentage of patients have positive for virus RNA by real time polymerase chain reaction(RT-PCR). | Up to Day 9
  The percentage of patients positive for virus RNA by RT-PCR.
The change from baseline in virus RNA by RT-PCR (unit: log₁₀ virus particles/mL). | Up to Day 9
  The change from baseline in the amount of virus RNA.
Area Under the Concentration (AUC) of virus RNA by RT-PCR and AUC of virus titer. | Up to Day 9
  AUC of the viral load by RT-PCR and AUC of viral titer measured from baseline to Day 9±2 or early termination (Visit 5).
The percentage of patients whose symptoms have been alleviated at each time point. | Up to Day 9
  The percentage of patients whose symptoms are alleviated at each time point.
The percentage of patients reporting normal temperature at each time point. | Up to Day 9
  The percentage of patients whose axillary temperature drops to less than 37ºC after the initiation of the study treatment in the analysis population.
Time to resolution of fever. | Up to Day 9
  The time between the initiation of the study treatment and the resolution of fever.
Body temperature at each time point. | Up to Day 9
  Measured axillary temperature.
Time to return to preinfluenza health status. | Up to Day 9
  Patients will be asked to record their pre-influenza health status between 0 (worst possible health) and 10 (normal health).
The visual analog scale (VAS) score change from baseline of quality of life (QOL) questionnaire. | Up to Day 9
  The VAS score change from baseline of QOL questionnaire.The QOL questionnaire consists 2 sections: the descriptive system and the VAS. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each of which is divided into 5 levels. The VAS records the patient's self-rated health on a 20-cm vertical visual analogue with "the best health the patient can imagine" as 100 and "the worst health the patient can imagine" as 0.
Incidence of influenza-related complications (hospitalization, death, sinusitis, bronchitis, otitis media, and radiologically confirmed pneumonia). | Up to Day 9
  The percentage of patients in the analysis population who experience each influenza-related complication (hospitalization, death, sinusitis, otitis media, bronchitis, and radiologically confirmed pneumonia) as an AE after the initiation of the study treatment.
The percentage of patients taking acetaminophen. | Up to Day 9
  The percentage of patients who took acetaminophen.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Huang, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Hunan, China